CLINICAL TRIAL: NCT01228890
Title: Primary Care Internet-Based Depression Prevention for Adolescents (CATCH-IT)
Acronym: CATCH-IT
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: no one enrolled; PI left institution
Sponsor: University of Chicago (Other)
Collaborators: Harvard Vanguard Medical Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-464-A
Record Dates: First submitted 2010-10-25; First posted 2010-10-27 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Depression; Anxiety; Externalizing Symptoms; Substance Abuse
MeSH Terms: conditions — Depression; Anxiety Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CATCH-IT 2-R Arm (Experimental): Primary care/Internet based depression prevention intervention (CATCH-IT 2-R) with a family component.
  Interventions: Behavioral: CATCH-IT
- Attention Monitoring Psycho-education (AMPE) Arm (Active Comparator)
  Interventions: Behavioral: AMPE

INTERVENTIONS:
Behavioral: CATCH-IT — The CATCH-IT 2-R intervention has a motivational (3 PCP motivational interviews at time 0, 1.5 months and 12 months and 3 coaching phone calls at 2 and 4 weeks and 18 months) and an Internet component (with separate adolescent [14 modules] and parent [5 modules] programs). This revised and expanded intervention will include a comprehensive approach to reducing modifiable risk factors and enhancing resiliency factors associated with increased or decreased risk of depression, respectively, proposed by Spence and Reinecke.148 The revised CATCH-IT "Tracker" will monitor time in study and deploy elements of the intervention based on time since enrollment, including computer and human elements (e.g. calls, doctor visits).
  Arms: CATCH-IT 2-R Arm
Behavioral: AMPE — The AMPE components are similar to those employed in previous primary care based quality improvement/Chronic Care Model Interventions (patient education [psycho-education described below], provider training [described in Case Finding and Recruitment], active monitoring and referral [case management, discussed under assessments], physician and nurse education and routine contact with PCP [study design rationale]). This Internet site will focus on assisting parents and adolescents in early identification of need for treatment and will also target stigma and negative attitudes toward treatment of mental disorders we have previously identified as barriers to seeking and adhering to treatment.
  Arms: Attention Monitoring Psycho-education (AMPE) Arm

SUMMARY:
In this 5-year, two-site randomized clinical trial, we propose to test the efficacy of the CATCH-IT primary care/Internet based depression prevention intervention against Attention Monitoring Psychoeducation (AMPE) in preventing the onset of depressive episodes in an intermediate to high risk group of adolescents aged 13-17. We plan to (a) identify high risk adolescents based on elevated scores on the PHQ-A, a screening measure of depressive symptoms; (b) recruit 400 (200 per site) of these at-risk adolescents to be randomized into either the CATCH-IT or the AMPE group; (c) assess outcomes at 2, 8, 12, 18, and 24 months post intake on measures of depressive symptoms, depressive diagnoses, other mental disorders, and on measures of role impairment in education, quality of life, attainment of educational milestones, and family functioning; and (d) conduct exploratory analyses to examine the effectiveness of this intervention program, moderators of protection, and potential ethnic and cultural differences in intervention response.

ELIGIBILITY:
Inclusion Criteria:

* Youth ages 13 through 17.
* Youth must be experiencing elevated level of depressive symptoms on the Center for Epidemiologic Studies Depression46 (CES-D) scale (score >/= 16) and have at least two core symptoms of Major Depression on the Patient Health Questionnaire, Adolescents.
* Youth will be included if they have a past history of depression, anxiety, externalizing symptoms, or substance abuse.

Exclusion Criteria:

* Current DSM-IV diagnosis (Kiddie Schedule of Affective Disorders) of Major Depressive Disorder, current therapy for depression, or be taking antidepressants (e.g., SSRIs, TCAs, MAOIs, bupropion, nefazodone, mirtazapine, venlafaxine).
* Current CES-D score >35
* DSM-IV diagnosis of schizophrenia (current or past) or bipolar affective disorder
* Current serious medical illness that causes significant disability or dysfunction
* Significant reading impairment (a minimum sixth-grade reading level based on parental report), mental retardation, or developmental disabilities
* Serious imminent suicidal risk (as determined by endorsement of current suicidality on CES-D or in KSADS interview) or other conditions that may require immediate psychiatric hospitalization
* Psychotic features or disorders, or currently be receiving psychotropic medication
* Extreme, current drug/alcohol abuse (greater than or equal to 2 on the CRAFFT).

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To determine whether the CATCH-IT 2-R depression prevention intervention prevents or delays major depressive episodes, as well as non-affective disorder episodes, compared to AMPE. | 49-60 months from beginning of trial

SECONDARY OUTCOMES:
To determine if participants in the CATCH-IT 2-R group exhibit more rapid favorable changes of depressive symptoms/and or vulnerability/protective factors compared with the AMPE group. | 49-60 months from beginning of the trial
To determine if participants in the CATCH-IT 2-R program report lower perceived educational impairment, greater quality of life, greater health-related quality of life, and lower incidence of other mental disorders (anxiety, substance/alcohol use). | 49-60 months from beginning of trial
To determine for whom (moderators) and how (mediators) the CATCH-IT 2-R program works in this population. | 49-60 months from beginning of trial

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Van Voorhees, MD, Principal Investigator — University of Chicago
Locations (4):
- United States (4):
  - University of Chicago, Chicago, Illinois
  - Access Community Health Network, Chicago, Illinois
  - Northshore University Health Systems, Evanston, Illinois
  - Harvard Vanguard Medical Associates, Boston, Massachusetts